CLINICAL TRIAL: NCT02101996
Title: Pilot Study to Test Dietary Fat Delivery
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Elizabeth Parks, Professor, University of Missouri-Columbia
Other Study IDs: 1211238
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Insulin Resistance
Keywords: stable isotopes; triacylglycerol
MeSH Terms: conditions — Insulin Resistance | interventions — Diet, High-Fat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and muscle biopsy samples are kept in Dr. Parks' lab for further study analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy: Not insulin resistant
  Interventions: Other: high-fat diet
- Insulin resistant: Insulin resistant by an insulin clamp
  Interventions: Other: high-fat diet

INTERVENTIONS:
Other: high-fat diet — Subjects consume a high-fat diet for three weeks before the in-hospital stay.

SUMMARY:
The average American diet consumed by a significant proportion of the adult population, supplies excessive calories and large amounts of saturated fat. Saturated fats can be cleared and used in skeletal muscle, but in obese individuals, biomarkers of saturated fat are found in the blood, along with markers of poor muscle metabolism.

Both fats and amino acids are processed by the same metabolic pathways in muscle, and the investigators hypothesize that meals with greater amounts of saturated fat slow muscle metabolism. A better understanding of the interaction of these to metabolites will allow for the development of future medications to treat muscle loss in sick individuals and the elderly.

DETAILED DESCRIPTION:
This study includes two parts, a baseline study and a three-week dietary study. The baseline study will be performed to test how the body absorbs and stores meal fat after a meal. In the three-week dietary study, the subjects will consume only the meals provided by the investigators for three weeks before the tests, and then participate in a hospital stay. The three-week dietary study is to test the chronic effect of a high fat diet on how body absorbs and stores the fat.

ELIGIBILITY:
Inclusion Criteria:

1. Lean/insulin sensitive (n=10, BMI ≤ 24 kg/m2 and glucose infusion > 4.0 mg/min))
2. Overweight/obese insulin resistant (n=10, BMI 26-35 and glucose infusion < 4.0 mg/min)
3. 30-50 years of age
4. Men and pre-menopausal women

Exclusion Criteria:

1. Insulin resistance is defined by insulin clamp as the rate of glucose infusion ≤ 4.0 mg/min.
2. BMI over 35 kg/m2
3. Abnormal thyroid function, kidney or liver disease
4. Uncontrolled hypertension, or occasional or regular smoker, use of medications or supplements that interfere with lipid, protein, or carbohydrate metabolism
5. Pregnancy (urine test), breast feeding an infant, or anemia
6. Alcohol intake: Males >140 g/week, Females > 70 g/week.
7. Fasting plasma triglycerides >300 mg/dL. Extreme hypertriglyceridemia could be due to either elevations in very low-density lipoproteins or chylomicrons, either of which would impair our ability to resolve dietary metabolic processes.
8. Need to consume acetaminophen-containing medications on a regular basis.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy and insulin resistant subjects.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-06; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Meal fat absorption and storage | Change in meal fat concentration in body tissues 8 h after two high-fat meals.
  Meal fat absorption and storage are measured using stable isotopes administration into sequential meals (breakfast and lunch). Analysis of plasma and muscle samples.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Parks, PhD, Principal Investigator — Univ of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

REFERENCES:
- [Background] Ramos-Roman MA, Sweetman L, Valdez MJ, Parks EJ. Postprandial changes in plasma acylcarnitine concentrations as markers of fatty acid flux in overweight and obesity. Metabolism. 2012 Feb;61(2):202-12. doi: 10.1016/j.metabol.2011.06.008. Epub 2011 Aug 5. PMID 21820684
- [Background] Ramos-Roman MA, Lapidot SA, Phair RD, Parks EJ. Insulin activation of plasma nonesterified fatty acid uptake in metabolic syndrome. Arterioscler Thromb Vasc Biol. 2012 Aug;32(8):1799-808. doi: 10.1161/ATVBAHA.112.250019. Epub 2012 Jun 21. PMID 22723441